CLINICAL TRIAL: NCT00018109
Title: A Multicenter Randomized Placebo-Controlled Double-Blind Study to Assess Efficacy and Safety of Glutamine and Creatine Monohydrate in Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's National Research Institute (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-5083
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Glutamine; Creatine

INTERVENTIONS:
Drug: glutamine
Drug: creatine monohydrate

SUMMARY:
To establish a collaborative group of clinical trial centers, with standardized equipment and protocols, able to conduct both drug and gene therapy trials in DMD. To evaluate the therapeutic effect of glutamine and creatine monohydrate on muscle strength in children with DMD. To validate the use of QMT (quantitative muscle strength testing) and gait analysis in children with DMD as reliable tools to quantify muscle strength, monitor disease progression and assess therapeutic response.

DETAILED DESCRIPTION:
Duchenne muscular dystrophy (DMD) is the most common lethal inherited disorder worldwide. Despite the exponential increase in our understanding of the disorder since the discovery and characterization of the causative gene and its product dystrophin in 1987, current therapeutic management remains largely supportive. Awaiting a final genetic cure to be available in the future, further investments in developing better drug therapies for DMD remain important. Not only because the uniform use of prednisone (the only drug proven to be beneficial) is hampered by potential adverse effects, but also because it may very well be the case that ultimately a combination of both gene and drug therapy will be needed to cure Duchenne children. Here, we test two compounds that have shown promise in a 45-drug screen in the mdx mouse model of Duchenne dystrophy.

The effect of glutamine (0.6/kg/day) and creatine monohydrate (5g/day) on muscle strength will be evaluated in a multi-center randomized double-blind placebo-controlled 3-arm study. Ambulant children aged 5-10 years with an established DMD diagnosis will be studied. Patients will undergo 2 screening evaluations within 2 weeks. Patients will be randomized into treatment groups on the second screening visits, followed by a 6-month treatment period. During the treatment period, patients will be evaluated at monthly intervals. The primary endpoints are percentage change in average muscle strength score and QMT performance for specific muscle groups. Secondary endpoints include timed function tests, functional grades for arms and legs, and pulmonary function tests.

ELIGIBILITY:
Ambulant children age 5-10 years with an established diagnosis of Duchenne Muscular Dystrophy

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States